CLINICAL TRIAL: NCT00118287
Title: Therapy of Myelodysplastic Syndrome (MDS) With Azacitidine Given in Combination With Etanercept: A Phase I/II Study.
Brief Title: Azacitidine and Etanercept in Treating Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bart Scott, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1926.00; NCI-2011-01818 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Secondary Myelodysplastic Syndromes
MeSH Terms: interventions — Azacitidine; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, chemoprotection) (Experimental): Patients receive etanercept SC twice weekly during weeks 1 and 2 and azacitidine SC or IV over 10-40 minutes on days 1-7. Treatment repeats every 28 days for at least 3 courses. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: azacitidine; Biological: etanercept

INTERVENTIONS:
Drug: azacitidine — Given SC or IV
  Other Names: 5-AC; 5-azacytidine; azacytidine; Vidaza
Biological: etanercept — Given SC
  Other Names: Enbrel; ETN; TNFR:Fc; Tumor Necrosis Factor Receptor IgG Chimera

SUMMARY:
This phase I/II trial studies how well giving azacitidine together with etanercept works in treating patients with myelodysplastic syndromes (MDS). Drugs used in chemotherapy, such as azacitidine, works in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Chemoprotective drugs, such as etanercept, may protect normal cells from the side effects of chemotherapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the frequency of hematologic responses in patients with MDS to 5-aza (azacitidine) plus etanercept.

II. Determine the efficacy of 5-aza combined with etanercept in patients with low or intermediate (int)-1 risk who fail to respond to anti-thymocyte globulin (ATG) plus etanercept and for the purpose of this trial are considered as having progressive or "more advanced" disease.

III. Correlate results of ex vivo/in vitro studies on phenotypic, cytogenetic and functional disease characteristics with in vivo treatment responses, to identify parameters that are associated with a high probability of response.

OUTLINE:

Patients receive etanercept subcutaneously (SC) twice weekly during weeks 1 and 2 and azacitidine SC or intravenously (IV) over 10-40 minutes on days 1-7. Treatment repeats every 28 days for at least 3 courses. Treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Int-2 or high risk MDS patients
* Patients with low-risk or int-1 risk MDS by International Prognostic Scoring System (IPSS) criteria with:

  * Single or multilineage cytopenia (absolute neutrophil count [ANC] < 1500/μL, hemoglobin [Hgb],10g/dL, or platelet count < 100,000/μL); or
  * Transfusion requirement of at least 2 units of packed red blood cells over an 8 week period
* Serum creatinine =< 1.5x ULN (upper limit of normal)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2x ULN
* Performance status =< 2 (Eastern Cooperative Oncology Group [ECOG] scale, 0-5)

Exclusion Criteria:

* Patients who have previously received hematopoietic stem cell transplants, specifically for MDS
* Patients with a diagnosis of acute myeloid leukemia (AML) by World Health Organization (WHO) criteria (i.e >= 20% blasts) at time of enrollment
* Women of child bearing potential who are currently pregnant, lactating or who are not willing to use contraception during the entire duration of the study
* Men who are unwilling to use contraception while receiving 5-aza
* Patients with severe disease other than MDS which is expected to prevent compliance with the present protocol
* Patients with severe infections (pneumonia, septicemia, etc) within the 2 weeks prior to the anticipated start of protocol treatment
* Patients who are currently receiving or within the preceding 2 weeks have received cytotoxic therapy, hemopoietic growth factors, immunomodulatory therapy, or other experimental therapy for the treatment of MDS
* Current evidence of uncontrolled cardiac arrhythmia or congestive heart failure
* Platelet count =< 10,000/mcl
* Absolute neutrophil count =< 250/mcl
* Prior treatment with 5-aza
* Known or suspected hypersensitivity to azacitidine or mannitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-04; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Scott, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Chemoprotection)
Started | 32
Completed | 30
Not Completed | 2
Not completed — Intracranial haemorrhage | 1
Not completed — Muscle pain | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Chemoprotection)
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 69 [31 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Hematologic Responses, as Defined by International Working Group (IWG) Criteria
Description: Count of participants with a hematologic improvement (erythroid, platelet, or neutrophil response), assessed at 3 months.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Chemoprotection)
Number analyzed (Participants) | 32
Participants
  Erythroid response | 14
  Platelet response | 8
  Neutrophil response | 1
  No response | 7
  Withdrawn from study | 2

ADVERSE EVENTS:
Arm/Group | Treatment (Chemotherapy, Chemoprotection)
Serious Adverse Events (participants affected / at risk) | 5/32
Other Adverse Events (participants affected / at risk) | 26/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Chemotherapy, Chemoprotection) (N=32)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Hemoptysis and fever (Respiratory, thoracic and mediastinal disorders) | 1
Cardiopulmonary arrest resulting in death (Cardiac disorders) | 1
Splenic rupture with splenectomy (Blood and lymphatic system disorders) | 1
Gall Bladder removal with benign mass (Hepatobiliary disorders) | 1
Pulmonary nodule (Respiratory, thoracic and mediastinal disorders) | 1
Endocarditis (Infections and infestations) | 1
CNS hemorrhages (Nervous system disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Chemotherapy, Chemoprotection) (N=32)
Anemia (Blood and lymphatic system disorders) | 19
Arthritis, Joint pain (Musculoskeletal and connective tissue disorders) | 5
Atrial fibrillation/flutter (Cardiac disorders) | 3
Bleeding from cuts (Skin and subcutaneous tissue disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6
Hematoma (Vascular disorders) | 2
Coagulopathy (Blood and lymphatic system disorders) | 3
Congestive heart failure (Cardiac disorders) | 6
Dehydration, 1 with diarrhea (Metabolism and nutrition disorders) | 2
Diverticulitis (Gastrointestinal disorders) | 2
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 3
Elevated cardiac enzymes (Cardiac disorders) | 3
Mouth/Gum Bleeding (General disorders) | 2
Fatigue (General disorders) | 11
Weakness (General disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Gallstones (Hepatobiliary disorders) | 2
Hematuria (Hepatobiliary disorders) | 9
Hives, urticaria (Skin and subcutaneous tissue disorders) | 3
Hyperbilirubinemia (Investigations) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7
Ileus (Gastrointestinal disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 15
Lymphopenia (Blood and lymphatic system disorders) | 16
Neutropenia (Investigations) | 17
Pleural effusions (Respiratory, thoracic and mediastinal disorders) | 2
Rectal or GI bleeding (Gastrointestinal disorders) | 6
Renal failure (Renal and urinary disorders) | 2
Thrombocytopenia (Investigations) | 17
Nausea/Vomiting (Gastrointestinal disorders) | 2
Compression fractures (Musculoskeletal and connective tissue disorders) | 2
Hypertension (Cardiac disorders) | 2
Squamos cell carcinoma removal (Skin and subcutaneous tissue disorders) | 2
Gout (Musculoskeletal and connective tissue disorders) | 2
Hypotension (Cardiac disorders) | 4
Transfusion reaction (Blood and lymphatic system disorders) | 3
Limited upper extremity function, after injury (Musculoskeletal and connective tissue disorders) | 2
Petechia (Blood and lymphatic system disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes